CLINICAL TRIAL: NCT06923969
Title: Effects of Balneotherapy on Echocardiographic Parameters in Adults and Elderly Patients With Osteoarthritis
Brief Title: Balneotherapy and Echocardiographic Findings in Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Taner Dandinoğlu, Physical Medicine and Rehabilitation (PM&R) physician, MD., Bursa City Hospital
Other Study IDs: 2026-PMR-6
Record Dates: First submitted 2025-03-23; First posted 2025-04-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis
Keywords: Balneotherapy; Echocardiography; Wellness; Heart
MeSH Terms: conditions — Osteoarthritis | interventions — Balneology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: balneotherapy

SUMMARY:
This prospective observational study aims to evaluate changes in heart function using echocardiography before and after a standardized balneotherapy program in adult and elderly patients with osteoarthritis.

Balneotherapy is commonly used by patients with osteoarthritis, especially in older age groups, who may also have known or unrecognized cardiovascular conditions. For this reason, heart function is evaluated using transthoracic echocardiography prior to the start of balneotherapy and again after completion of the treatment program.

The study focuses on changes in echocardiographic parameters related to left ventricular systolic and diastolic function. By comparing measurements obtained before and after balneotherapy, this study seeks to improve understanding of the potential effects of balneotherapy on cardiac function in patients with osteoarthritis.

DETAILED DESCRIPTION:
Balneotherapy is frequently preferred by adult and elderly patients with osteoarthritis as part of rehabilitation programs. This population may have a higher prevalence of overt or subclinical cardiovascular disease; therefore, cardiovascular evaluation before and after balneotherapy may be clinically relevant.

In this prospective observational study, patients with osteoarthritis who are scheduled to undergo a standardized balneotherapy program are evaluated using transthoracic echocardiography prior to treatment initiation and again after completion of the program. Echocardiographic examinations are performed to assess parameters related to left ventricular systolic and diastolic function, as well as aortic hemodynamics.

The balneotherapy program consists of head-out immersion in thermal pools with acratothermal water at a temperature of approximately 38 °C, applied for 20 minutes per session, 5 days per week, over a 15-day period. Echocardiographic measurements obtained before and after the intervention are compared to evaluate potential changes in cardiac function associated with balneotherapy.

ELIGIBILITY:
Inclusion Criterias:

* Having balneotherapy sessions 5 days a week for total of three weeks
* Having detailed echocardiography records

Exclusion Criterias:

* Having history of major surgery,
* cerebrovascular accident,
* malignancy,
* liver or renal failure,
* immunodeficiency,
* acute/chronic infection,
* psychiatric disorders were exluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult and elderly patients diagnosed with osteoarthritis who are scheduled to undergo a standardized balneotherapy program at a tertiary care rehabilitation hospital. Eligible participants undergo transthoracic echocardiographic evaluation before initiation of balneotherapy and again after completion of the treatment program in order to assess potential changes in cardiac function.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Change in mitral peak E wave velocity | Baseline (before balneotherapy) and immediately after completion of the 15-day balneotherapy program
  Change in mitral peak early diastolic (E) wave velocity measured by transthoracic echocardiography.
Change in mitral E/A ratio | Baseline and immediately after completion of the 15-day balneotherapy program
  Change in the ratio of early (E) to late (A) diastolic transmitral flow velocities assessed by transthoracic echocardiography.
Change in E/E' ratio | Baseline and immediately after completion of the 15-day balneotherapy program
  Change in the ratio of early transmitral flow velocity (E) to early diastolic mitral annular velocity (E') measured by tissue Doppler imaging.

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction | Baseline (before balneotherapy) and immediately after completion of the 15-day balneotherapy program
  Change in left ventricular ejection fraction assessed by transthoracic echocardiography.
Change in mean aortic gradient | Baseline (before balneotherapy) and immediately after completion of the 15-day balneotherapy program
  Change in mean transaortic pressure gradient measured by continuous-wave Doppler echocardiography.
Change in maximum aortic gradient | Baseline (before balneotherapy) and immediately after completion of the 15-day balneotherapy program
  Change in maximum transaortic pressure gradient measured by continuous-wave Doppler echocardiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Military Hospital, 1. Murat Caddesi Osmangazi, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Research data will be available upon request from author
  (Taner Dandinoglu MD. e-mail: dandinoglu@gmail.com)